CLINICAL TRIAL: NCT07108777
Title: Clinical Study to Evaluate the Possible Protective Effect of L-Carnitine Against Cisplatin-Induced Nephrotoxicity
Brief Title: L-Carnitine Protective Effect in Nephrotoxicity
Acronym: LC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Fatma Mamdouh Elsayed Eweda, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ONCO21
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Nephrotoxicity
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-carnitine group (Active Comparator): This group will receive the standard chemotherapy protocol (cisplatin -based chemotherapy) plus L-carnitine 350 mg (L-carnitine®) three times daily by oral.
  Interventions: Drug: L-Carnitine Tartrate
- Placebo group (Placebo Comparator): This group will receive the standard chemotherapy protocol (cisplatin -based chemotherapy) plus placebo tablets with the same criteria of the intervention drug and the same dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Carnitine Tartrate — L-carnitine 350 mg three times daily by oral.
  Other Names: L-Carnitine, Levocarnitine, carnitine
  Arms: L-carnitine group
Drug: Placebo — placebo tablet three times daily by oral.
  Other Names: Matching placebo, inactive control
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to assess the possible reno-protective effect of L-carnitine against cisplatin-induced nephrotoxicity in patients receiving cisplatin-based chemotherapy. The main question it aims to answer is:

Does L-carnitine have the ability to protect the kidney against cisplatin-induced nephrotoxicity?

DETAILED DESCRIPTION:
Cisplatin is one of the most effective chemotherapeutic agents that has been used for more than 50 years for a different solid Tumers. Nevertheless, its administration is associated with toxicity, including nephrotoxicity which can affects 25-35% of treated patients. Cisplatin nephrotoxicity mainly explained by accumulation in the renal tubules mostly in the proximal and distal tubules where it inhibits and alters the expression pattern of several membrane transporters and water channels and inhibits mitochondrial function and ATP production, thus generating oxidative stress. Cisplatin nephrotoxicity is also associated with an inflammatory response that plays a significant role in this event. Tumor necrosis factor alpha (TNF- α) is a pleiotropic pro-inflammatory cytokine that signals via TNFRSF1A and TNFRSF1B to activate nuclear factor kappa B (NF-κB) or Mitogen-activated protein kinase (MAPK), eventually leading to cytokine production and/or death signaling. L-carnitine owing to its antioxidant and anti-inflammatory properties has been used as a candidate for nephroprotection against drug induced nephrotoxicity (DIN). L-carnitine significantly ameliorates DIN in animal studies especially against cisplatin-induced renal damage. Inhibition of reactive oxygen species generation, lipid peroxidation, matrix remodeling and apoptosis, anti-inflammatory properties and improvement in carnitine deficiency has been suggested as probable nephroprotective mechanisms of L-carnitine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients.
* Newly diagnosed patients with cancer and with an indication for cisplatin - based chemotherapy.
* Age between 18 and 75 years.
* No serious cardiopulmonary comorbidity which could impair involvement in the study.
* Creatinine clearance value above 50 mL/min/1.73 m².
* Patients who will scheduled to receive at least 3 cycles of cisplatin.
* Patients with no previous renal diseases (including acute nephropathy, acute and chronic renal failure).

Exclusion Criteria:

* Pregnancy or lactation.
* Metastasis to the central nervous system.
* Psychiatric disorders.
* Prior treatment with platinum derivatives.
* Hypersensitivity to cisplatin, carboplatin or other platinum derivatives.
* Patients with active infection or any symptoms of sepsis.
* Acute renal failure or renal surgery within the last 3 months.
* Patients unfit for cisplatin (patients with impaired renal function, sensorineural hearing loss and cardiomyopathy).
* Patients with known history or current treatment with nephrotoxic agents.
* Taking other antioxidant supplements such as Vitamins C and E.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
change in serum creatinine and creatinine clearance | Baseline (before chemotherapy cycles)
  serum creatinine average ranges are 0.7 to 1.2 (mg/dL) for males and 0.5 to 1.0 for females.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma M Eweda, Master, Principal Investigator — Tanta University
Locations (1):
- Menoufia Clinical Oncology Department, Menoufia University., Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No